CLINICAL TRIAL: NCT05130619
Title: Human Auto-ethanol Formation and Acetate Signaling. Acute Effects of Alcohol on Short-chain Fatty Acid Dynamics and Energy Metabolism in Healthy Men and Women.
Brief Title: Human Auto-ethanol Formation and Acetate Signaling
Acronym: HotFacets
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Copenhagen (Other)
Responsible Party: Principal Investigator, Professor Lars Ove Dragsted, Professor, University of Copenhagen
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Basic Science
Other Study IDs: M240
Record Dates: First submitted 2021-10-14; First posted 2021-11-23 (Actual); Last update posted 2023-11-30 (Actual); Status verified 2023-11

CONDITIONS: Healthy
MeSH Terms: interventions — Ethanol

STUDY DESIGN:
Who Masked: Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Treatment order A-.B-C-D (Experimental): A: 5g ethanol-2-D3 mixed into 250ml water with added aromas of gin and lime juice B:10g ethanol-2-D3 mixed into 250ml water with added aromas of gin and lime juice C: 8g Triacetin mixed into 250ml water with added aromas of gin and lime juice D: 250ml water with added aromas of gin and lime juice
  Interventions: Dietary Supplement: Ethanol
- Treatment order B-D-A-C (Experimental): A: 5g ethanol-2-D3 mixed into 250ml water with added aromas of gin and lime juice B:10g ethanol-2-D3 mixed into 250ml water with added aromas of gin and lime juice C: 8g Triacetin mixed into 250ml water with added aromas of gin and lime juice D: 250ml water with added aromas of gin and lime juice
  Interventions: Dietary Supplement: Ethanol
- Treatment order C-A-D-B (Experimental): A: 5g ethanol-2-D3 mixed into 250ml water with added aromas of gin and lime juice B:10g ethanol-2-D3 mixed into 250ml water with added aromas of gin and lime juice C: 8g Triacetin mixed into 250ml water with added aromas of gin and lime juice D: 250ml water with added aromas of gin and lime juice
  Interventions: Dietary Supplement: Ethanol
- Treatment order D-C-B-A (Experimental): A: 5g ethanol-2-D3 mixed into 250ml water with added aromas of gin and lime juice B:10g ethanol-2-D3 mixed into 250ml water with added aromas of gin and lime juice C: 8g Triacetin mixed into 250ml water with added aromas of gin and lime juice D: 250ml water with added aromas of gin and lime juice
  Interventions: Dietary Supplement: Ethanol

INTERVENTIONS:
Dietary Supplement: Ethanol — Crossover meal study

SUMMARY:
The HotFacets study is a randomized, controlled, cross-over meal study that investigates the acute effects of alcohol consumption on short-chain fatty acids dynamics, energy metabolism, and biomarkers.

Despite the negative health consequences of chronic alcohol abuse, observational and cohort studies associate moderate alcohol consumption with a 20-30 % lower risk of cardiovascular diseases (CVD) and Type 2 Diabetes Mellitus (T2DM), compared to abstainers. Based on the J-shaped relationship between alcohol intake and the risk of cardiometabolic diseases, ½-2 standard drinks/day can be considered as moderate alcohol consumption. The interpretation of the J-shaped relationship has been criticized mainly due to potential confounding from the selected reference group and uncontrolled lifestyle factors. Longer, well-designed randomized controlled trials are lacking to infer causality and to clarify the mechanism of action for the acute and chronic effects of moderate alcohol consumption on cardiometabolic health and energy homeostasis. However, some aspects of alcohol metabolism and biomarker validation could inform such a study.

HotFacets is set to generate insight into the effects of acute alcohol intake on SCFA dynamics in blood, urine, and faeces; into the dose-response relationship with REE, thermogenesis, substrate oxidation, and alcohol biomarkers; and to explore potential low levels of alcohol produced in the gut.

DETAILED DESCRIPTION:
A randomized, controlled, four times cross-over, single-blinded, meal study with 24 healthy fasting subjects will be conducted with a) placebo (water), b) a metabolic acetate generator (triacetin), and c) a half or d) one unit of isotope labelled ethanol, provided in a randomized order. Volunteers will be confined in a metabolic chamber overnight before each test drink (in 250mL water with lemon and juniper taste) and energy production and expenditure will be measured initially using seven ventilated hood measurements. After the test drinks and ventilated hood measurements an ad libitum lunch will be served before the participants will be admitted to the metabolic chamber, where metabolic measurements will be continued until the following day. Participants will go through a 2-week run-in period before each test drink and a 2-week wash out period afterwards, both with alcohol abstention. From two days before the test day in each period until one day after the test days, standardized foods will be provided. Anthropometrics, DXA, heart rate, blood pressure and all movements will be recorded before and/or during the test days. Before, during, and after the test day repeated biological samples (i.e., urine, blood, feces, hair) will be collected. The study will be divided into a pre-trial (8 subjects, 50-75y) and a main trial (16 subjects, 25-75y).

ELIGIBILITY:
Subjects will be recruited to the trial in two seasons. First, eight healthy men and post-menopausal women 50-75 years will be recruited for the pre-trial during autumn/winter 2021. Secondly, 16 healthy men and women with an age-range of 25-75 years will be recruited for the main trial during late spring/summer 2022.

Age-specific inclusion criteria for the pre-trial:

* Healthy men and healthy, post-menopausal women (12 consecutive months without menstrual period)
* Age: 50-75 years old
* BP ≤ 140/90 (systolic/diastolic)
* Plasma glucose <7 mmol/l
* BMI: 18.5-27 kg/m2
* Subjects with a good command of both written and verbal English

Age-specific inclusion criteria for the main-trial:

* Healthy men and women
* Age: 25-75 years old
* BP ≤ 140/90 (systolic/diastolic)
* Plasma glucose <7 mmol/l
* BMI: 18.5-27 kg/m2

Inclusion criteria for the pre- and main-trial:

* Willing to provide registration of compliance during the run-in period and follow-up periods
* Willing to avoid drinking alcohol for 2 weeks before the first test day and between test days
* Willing to stay in the respiration chamber the night before and after each test day
* Owning a smartphone

Exclusion Criteria:

* Alcohol naïve or has not consumed alcohol within the last year
* Any history of alcohol or substance abuse or a high alcohol intake, defined as:

  * An Alcohol Use Disorders Identification Test (AUDIT, appendix 1) score > 5 at screening
  * Drinking on average >14 alcoholic beverages a week during the past 6 months
  * Yale-Brown Obsessive Compulsive Scale-heavy drinking (Y-BOCS-hd, appendix 2) total score of ≥6 on questions 1, 2, and 3
* Intolerance or allergy to alcoholic beverages, juniper or citrus
* Diagnosed with any CVD event (MI, revascularization procedure or stroke) within the past six months
* Diagnosed with any known or past severe chronic disease including liver diseases (e.g., active hepatitis B and C infections, liver cirrhosis, hepatitis, cancer), T2DM, prediabetes, hypertension, severe psychiatric illness or frequent use of medication (except over-the-counter drugs or mild anti-depressants) or any other clinical condition that makes the subject ineligible according to the clinically responsible medical doctor (self-reported).
* Cancer - active malignant cancer or history of malignancy within the last 5 years (with exception of non-melanoma skin cancer).
* Previous breast cancer diagnosis or at high risk of breast cancer defined as:

  * Breast Cancer Risk Assessment Tool (BCRAT) risk score > 5 % (https://bcrisktool.cancer.gov/calculator.html)
  * Close relatives with diagnosed breast cancer (mother, sister, daughter)
* A Patient Health Questionnaire (PHQ-9, appendix 3) ≥15 at screening or a positive response on question 9 (thoughts about suicide)
* Diagnosed with atrial fibrillation
* Hemoglobin (Hb) levels below 7.3 mmol/L for women and 8.3 mmol/L for men.
* Chronic use of any type of medication, except for mild antidepressants or contraceptives
* Any use of contraindicated medication for alcohol intake, such as disulfiram, dual antiplatelet therapy, metronidazole, warfarin or hormone replacement therapy
* Hypersensitive to plasters
* Use of any type of antibiotics within two month before the first test day
* Unintentional weight loss >20% during the last 6 months
* Any type of gastrointestinal problems or prior surgery expected to influence gut health and absorption.
* Estimated glomerular filtration rate (eGFR) < 30 ml/min/1.73 m2 or end-stage renal disease
* Liver function tests >2 times the upper limit of the normal range according to current limits at "sundhed.dk": alanine transaminase (ALT), aspartate aminotransferase (AST), and gamma-glutamyltransferase (GGT).
* Blood donations within the past three months before the recruitment
* Having no hair on the head (bald-headed)
* Current participation in another trial
* Not willing to sign the Informed consent form (ICF)
* Not willing to comply with the all the trial procedures including completion of the two-week run-in periods without drinking alcohol as well the two-week wash-out periods
* Unable or unwilling to follow the safety procedures related to Covid19
* Any other issue that makes the project responsible researcher doubt the eligibility of the volunteer

Ages: 25 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 24 (Estimated)
Dates: Start 2021-11-10 (Actual); Primary Completion 2024-04-01 (Estimated); Study Completion 2024-12 (Estimated)

PRIMARY OUTCOMES:
SCFA dynamics | 0-48 hours after intake
  Difference in isotope labelled and unlabelled SCFA (mainly acetate, butyrate and propionate) concentration time course in feces, blood and urine following one unit of alcohol intake compared with half a unit, triacetin or water.

SECONDARY OUTCOMES:
Resting energy expenditure | 0-3 hours after intake
  Difference in resting energy expenditure, diet induced thermogenesis, and substrate oxidation following one unit of alcohol intake compared with half a unit, triacetin or water.
substrate oxidation rate | 0-3 hours after intake
  Difference in resting energy expenditure, diet induced thermogenesis, and substrate oxidation following one unit of alcohol intake compared with half a unit, triacetin or water.
diet induced thermogenesis | 0-3 hours after intake
  Difference in resting energy expenditure, diet induced thermogenesis, and substrate oxidation following one unit of alcohol intake compared with half a unit, triacetin or water.
Biomarkers of alcohol intake in hair | 0-1 month after intake
  Difference in alcohol biomarker levels of ethyl glucuronide, ethyl sulphate and fatty acid ethyl esters in hair following one unit of alcohol intake compared with half a unit, triacetin or water.
Biomarkers of alcohol intake in urine | 0-1 month after intake
  Difference in alcohol biomarker levels in urine following one unit of alcohol intake compared with half a unit, triacetin or water.
Biomarkers of alcohol intake in red blood cells | 0-1 month after intake
  Difference in alcohol biomarker levels in red blood cells following one unit of alcohol intake compared with half a unit, triacetin or water.
Biomarkers of alcohol intake in blood serum or plasma | 0-1 month after intake
  Difference in alcohol biomarker levels in blood serum or plasma following one unit of alcohol intake compared with half a unit, triacetin or water.
Low-level endogenous alcohol production measured as biomarkers of ethanol exposure during strict abstention in a metabolic chamber | 0-48 hours after intake
  Difference in low-level baseline alcohol production by the yeast and bacteria in the gut following one unit of alcohol intake compared with half a unit, triacetin or water.
Isotope labelled metabolites | 0-48 hours after intake
  Difference in metabolites of (non-radioactive) isotope-labelled ethanol compared with triacetin ingestion in blood, red blood cells, urine, faeces and hair; these metabolites are measured by liquid chromatography time-of-flight mass spectrometry as an increase in the third isotope peak for any molecular mass feature in the chromatogram.
Heart rate and blood pressure | 0-24 hours after intake
  Difference in heart rate and BP including diurnal biphasic systolic and diastolic fluctuations measured through 24-hour ambulatory BP after one unit of alcohol intake compared with half a unit, triacetin or water.
Alcohol levels in breath | 0-8 hours after intake
  Difference in alcohol levels measured by an alcohol breath analyzer after one unit of alcohol intake compared with half a unit, triacetin or water.

OTHER OUTCOMES:
Microbiome composition | 0-48 hours after intake
  Differences in taxonomic composition (relative or absolute) of the gut microbiota when comparing one unit of alcohol intake compared with half a unit, triacetin or water.
Microbiome functionality | 0-48 hours after intake
  Differences in alcohol-producing functional composition of the oral and gut microbiota, when comparing samples collected before and after one unit of alcohol intake compared with half a unit, triacetin or water. This fundtional composition is determined by the relative abundance of Anaerostipes caccae, Bacteroides thetaiotaomicron, Bifidobacterium longum, Enterococcus fecalis, Escherichia coli, Lactobacillus acidophilus, Lactobacillus fermentum, Lactobacillus plantarum, Weissella confusa, Clostridium subclusters IV and XIVa, Saccharomyces cerevisiae, Candida albicans and any other established alcohol-producing microbiota.
Faecal pH | 0-48 hours after intake
  Differences in faecal pH, when comparing one unit of alcohol intake compared with half a unit, triacetin or water.
Metabolic fingerprints of urine | 0-48 hours after intake
  Difference in metabolomes of urine when comparing samples taken up to 48 hours after one unit of alcohol intake compared with half a unit, triacetin or water. The LC-MS and NMR metabolomes will be compared by PLS-DA to find discriminant patterns of metabolic features.
Metabolic fingerprints of plasma or serum | 0-48 hours after intake
  Difference in metabolomes of blood serum/plasma when comparing samples collected after one unit of alcohol intake compared with half a unit, triacetin or water. The LC-MS and NMR metabolomes will be compared by PLS-DA to find discriminant patterns of metabolic features.
Metabolic fingerprints of feces | 0-48 hours after intake
  Difference in metabolomes of feces, when comparing samples collected after one unit of alcohol intake compared with half a unit, triacetin or water. The LC-MS and NMR metabolomes will be compared by PLS-DA to find discriminant patterns of metabolic features.

CONTACTS AND LOCATIONS:
Overall Officials: Lars O Dragsted, PhD, Principal Investigator — University of Copenhagen
Locations (2):
- Denmark (2):
  - Department of Nutrition, Exercise and Sports, University of Copenhagen, Copenhagen, Frederiksberg C
  - Lars Ove Dragsted, Frederiksberg

IPD SHARING:
Plan to Share IPD: No
Samples are to be anonymized before being shared with other researchers if the case.